CLINICAL TRIAL: NCT02621788
Title: Evaluation of Mind-body Educational Program to Enhance Resiliency and Reduce Burnout in First Year Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Director of Research, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000234
Record Dates: First submitted 2015-05-14; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Stress
Keywords: mind/body medicine; 3RP; stress management; resident burnout

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- First Year Residents (Experimental): Stress Management and Resiliency Training for Residents (SMART-R) delivered to first year residents in the departments of medicine and psychiatry at Massachusetts General Hospital
  Interventions: Behavioral: Stress Management and Resiliency Training for Residents (SMART-R)

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training for Residents (SMART-R) — The SMART-R is a mind-body Educational Program for residents that is aimed at reducing the impact of stress and enhancing coping strategies through skill building exercises. The intervention consists of 3, 2 hour sessions over the course of 12 months.

SUMMARY:
This prospective pilot study evaluated the benefits of a stress management and resiliency training program for residents (SMART-R).

The primary objective of this study is to determine whether the SMART-R effectively reduces burnout and stress and enhances coping skills in first year residents. Objective parameters (heart rate, galvanized skin response, sleep duration and quality, exercise and actigraphy) measured with the Basis health tracking device will help correlate objective signs to subjective report of stress.

The investigators' hypothesis is that the SMART-R, a curriculum designed to teach first year residents (in the department of Medicine and Psychiatry) relaxation skills, will enhance residents' emotional and physical well being, reduce reports of stress, anxiety, depression, and physical complaints, as well as increase overall resiliency.

DETAILED DESCRIPTION:
The SMART-R has been developed by the Benson-Henry Institute (BHI) of Mind Body Medicine and is aimed at reducing the impact of stress through a variety of skill building exercises. The exercises incorporated into the program have been shown to improve physical symptoms, mood and wellbeing in medical patient populations. However, very little work has focused on healthcare providers, and there are no studies that look at mindfulness interventions for resident physicians specifically.

Participants enrolled will be invited to complete a set of questionnaire before and after participation in the program. The investigators will also collect continuous physiologic data using the Basis Peak Health Tracking device to correlate the physiologic data with self-report measures of stress.

ELIGIBILITY:
Inclusion Criteria:

* Massachusetts General Hospital first year resident in Department of Medicine or Department of Psychiatry
* 21 years of age or older
* consenting to participate in 3RP-1

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in burnout levels post intervention | change between baseline (week 0) and post intervention (week 52)
  Maslach Burnout Inventory (MBI), a validated 22-item self-report measure of professional burnout in human services. The MBI consists of 3 subscales of burnout: emotional exhaustion, depersonalization, and low sense of personal accomplishment.
Change in perceived stress post intervention | change between baseline (week 0) and post intervention (week 52)
  Perceived Stress Scale (PSS-10)
Change in continuous physiologic data throughout intervention | change between baseline (week 0) and post intervention (week 52)
  Basis Peak Health Tracking device collects continuous physiologic data (heart rate, galvanized skin response, sleep duration and quality, exercise and actigraphy)
change in coping abilities post intervention | change between baseline (week 0) and post intervention (week 52)
  Measure of Coping Status-Revised (MOCS-R)

SECONDARY OUTCOMES:
change in self-reported anxiety and depression | change between baseline (week 0) and post intervention (week 52)
  Beck Anxiety Inventory (BAI) and Patient Health Questionnaire 9-item

CONTACTS AND LOCATIONS:
Overall Officials: John Denninger, M.D./PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH department of medicine and department of psychiatry, Boston, Massachusetts, United States